CLINICAL TRIAL: NCT06157814
Title: Mobile Ostomates Resources Intervention for Patients and Caregivers
Brief Title: Mobile Ostomates Resources for Patients and Caregivers
Acronym: MORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Nihal E Mohamed, Associate Professor of Urology, Director of Patient Education & Behavioral Research, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY-22-00556
Record Dates: First submitted 2023-08-08; First posted 2023-12-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Colorectal Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients recruited, aside from their caregivers, will have already received OR are scheduled for ostomy surgery. Patient and caregivers will be randomized 1:1 to the control and intervention group. The intervention group of patents and caregivers will be given access to the STOMA Care app while the control group of patents and caregivers will NOT be given access to the STOMA Care app during the course of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STOMA Care (Experimental): Patients and the caregivers accessing the full MORE program on the secured Website. The patients and caregivers will be instructed on how to complete the 1 week (or upon discharge) and 4 week surveys via REDCap or through the RC. This group has additional requirements in the 4-week survey to assess the helpfulness of the Stoma Care app.
  Interventions: Other: STOMA Care web-based application
- Usual Care (Active Comparator): Patients and caregivers will NOT be given access to the web-based app and outpatient clinic will provide ostomy care if requested by all patients with ostomies per their regular care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: STOMA Care web-based application — The STOMA Care App, with program software developed in collaboration with the Information Technology Department at Mount Sinai, is organized in a web-based app accessible on any smart-phone (e.g., Android and iOS), tablet, or computer device and consist of: 1) provision of information through text, and graphics; 2) videos of physicians and nurses answering questions; and 3) videos of patients describing their experiences and modelling competencies 4) mental health, support group, and ostomy supplier resources.
  Other Names: STOMA Care
  Arms: STOMA Care
Other: Usual Care — Patients and caregivers NOT given access to the web-based application.
  Arms: Usual Care

SUMMARY:
The scope of this research is to examine the acceptability and feasibility of a refined web-based intervention ("STOMA Care" app) by conducting a randomized pilot consisting of bladder and colorectal cancer patients scheduled for ostomy surgery at Mount Sinai Health System and their primary caregivers. This study aims to explore the impact of the app on stoma-related knowledge and beliefs, patient stoma-care skills and self-efficacy beliefs, and self-regulation and adaptation (e.g., distress and quality of life) among patients and their informal caregivers.

DETAILED DESCRIPTION:
The MORE study was designed guided by the Individual and Family Self-Management Theory to facilitate adaptation to stoma care within three key patient and caregiver unmet need domains: 1) enhancement of knowledge and beliefs (e.g., outcome expectations), 2) enhancement of ostomy-care competencies (e.g., learning skills and building confidence), and 3) enhancement of self-regulation (e.g., stress management). Content for these domains is organized in a web-based app (STOMA Care) accessible on any smart-phone (e.g., Android and iOS), tablet, or computer device and consist of: 1) provision of information through text, and graphics; 2) videos of physicians and nurses answering questions; and 3) videos of patients describing their experiences and modeling competencies. Program software was developed in collaboration with the Information Technology Department at Mount Sinai. A usability testing with 11 patients, caregivers, and nurses showed high acceptability and usability of MORE and led to refinements of the program software. In this proposed pilot study, the research team plan to examine the acceptability and feasibility of the refined MORE in bladder and colorectal cancer patients with new ostomies and their family caregivers. Results from this pilot study will inform a large randomized clinical trial (RCT) of MORE with ostomy patients and their caregivers. Here researchers aim to: Aim 1: Examine the acceptability and feasibility of the refined MORE: The research team will conduct a pilot, randomized, feasibility study with 45 bladder and colorectal cancer patients scheduled for ostomies at Mount Sinai Health System and their family caregivers. The primary outcomes of interest will be measures of feasibility and acceptability of MORE. Feasibility will be evaluated based on the ability to recruit and randomize participants (patient/caregiver dyads) to the two treatment arms (MORE vs. usual care), retain participants for the entire duration of the study period, apply appropriate methods for assessment and implement the program in a diverse, urban ostomy patient population and their family caregivers. Pre- and post-surgical secondary outcomes measured by standardized scales (1 week before surgery; day of discharge, and 4 weeks post-discharge) for the following variables will be used to estimate effect size for powering a larger future RCT: stoma-related knowledge and beliefs, patient stoma-care skills and self-efficacy beliefs, and self-regulation and adaptation (e.g., distress and quality of life). The research team hypothesize that MORE will be acceptable and feasible, will improve patient and caregiver knowledge, stoma-care skills, and quality of life, and will reduce their emotional distress.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ostomy surgeries for bladder or colorectal cancer;
* Age 21 or older
* Physically and mentally able to consent and participate
* Access to a phone
* Able to speak/read/write English
* Has an informal/family caregiver (age 21 or greater) willing to participate in the study

Exclusion Criteria:

* Patients with metastatic cancer, cancer recurrence, or presence of other cancers
* Not able to speak/read/write English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | Duration of study (5 weeks)
  Feasibility will be evaluated based on the research team's ability to recruit participants.
Number of participants retained for entirety of the study | Duration of study (5 weeks)
  Feasibility will be evaluated based on the research team's ability to recruit participants retain participants for the entire duration of the study period, apply appropriate methods for assessment and implement the program in a diverse, urban ostomy patient population and their family caregivers.

SECONDARY OUTCOMES:
Stoma/Ostomy Knowledge Questionnaire | Duration of study (5 weeks)
  This questionnaire assesses respondents' knowledge of standard ostomy care procedures (reaction to stoma, removing the stoma appliance, measuring the stoma diameter, adjusting the size of the stoma diameter in a new stoma appliance, skin care, fitting a new stoma appliance, and emptying procedure). Minimum score = 0, Maximum score = 21. A higher score indicates higher skill in ostomy care with less dependence on an ostomy nurse.
Illness Perception Questionnaire (IPQ) | Duration of study (5 weeks)
  This questionnaire assesses five cognitive illnesses. Responses to the items can be grouped into categories such as stress, lifestyle, etc. to measure respondents' perception of illness. Subscale scores range from 1-10. Minimum score= 0, Maximum score= 80; higher scores indicate worse illness perception.
  Eight items in addition to a causal scale graded on a five-point Likert scale.
The General Self-Efficacy Scale | Duration of study (5 weeks)
  This scale assesses a general sense of perceived self-efficacy, predicting respondents' ability to cope with daily hassles and adaptation after stressful life events. Minimum score = 10, Maximum score = 40; higher scores indicate higher self-efficacy.
Adapted Quality of Life Questionnaire for Patients with an Ostomy | Duration of study (5 weeks)
  Questions adopted from the Quality-of-Life Scale, respondents will elaborate on their difficulties in stoma care, surgery and treatment-related goals, then indicate whether they have achieved their goals and how satisfied they are with their achievement. For each item, 0 = worst outcome/negative QOL and 10 = best outcome/positive QOL. A total QOL score is obtained by adding the scores on all 10-point items and dividing by the total number of items (43). Minimum score = 0, Maximum score = 10. Higher scores indicate a general better quality of life among ostomates.
Number of nurse home visits | Duration of study (5 weeks)
Number of visits to emergency room | Duration of study (5 weeks)
Brief Symptoms Inventory (BSI-18) Score | Duration of study (5 weeks)
  Brief Symptoms Inventory (BSI-18) will measure respondents' distress symptoms. The assessment contains three six-item scales for measuring somatization, depression, anxiety, and the Global Severity Index (GSI). Respondents rate items on a scale from "Not at all," indicating low psychological distress, to "Extremely," indicating high psychological distress in that area. Thus, higher responses of "Extremely" across the scales signify greater distress in that area being measured. Subscale scores range from 1-5. Minimum score = 0, Maximum score = 90; higher scores indicate more distress.
Quality of Life Questionnaire for Patients with an Ostomy | Duration of study (5 weeks)
  This 43-item scale assesses the psychological, social, and spiritual wellbeing of respondents, graded on a 0-10 scale in which 0 reflects very poor quality in that area and 10 is the best. Total quality of life (QOL) is calculated by adding the scores on all of the 10-point items. Minimum score = 0, maximum = 430. Higher scores indicate a better quality of life.
Unmet Needs | Duration of study (5 weeks)
  This measure assesses respondents' needs including psychological, physical, informational, daily living, patient care, and sexuality needs. Respondents may choose one of five possible responses to all 33 questions ranging from "No need" to High need". Minimum score = 1, Maximum score = 165. Higher need answers indicate greater unmet needs.
Satisfaction with Care/Communication | Duration of study (5 weeks)
  This measure assesses satisfaction with care and communication between cancer in patients with hospital-based care and their care team, caretakers, and significant others. Respondent's report how much each of 11 statements apply to them within the past month using the five responses ranging from "Not much" to "Very much". Minimum score = 1, Maximum score = 55. Higher responses of "very much" indicate low satisfaction.
Symptom Measures | Duration of study (5 weeks)
  Symptoms of pain, fatigue, anxiety, and depression will be reported as a composite score, measured using five questions with scales ranging from 0 (none) to 10 (the worst imaginable) as well as the impact that these symptoms have on respondents' quality of life measured using three questions with scales ranging from 1(none) to 5 (very great impact. Full composite score from 5 to 40 A higher score indicates more adverse physical and psychological symptoms experienced and poorer quality of life as a result of the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Mohamed, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to being used to complete this research study, personal information (such as, name, address, date of birth, social security number), study data, may also be used and shared for additional (future) research. Before anything is shared, identifying personal information will be removed and it will be replaced with a code. Researchers are not planning on giving you the details of any of this future research nor the results. If patients do not want any future research to be done with your data and/or samples, even with identity removed, they will not be included in this study.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available after ICF is signed and will be available and does not expire.